CLINICAL TRIAL: NCT02114606
Title: Diagnosis and Monitoring of Eosinophilic Esophagitis Using the Cytosponge
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Cytosponge device availability
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Mayo Clinic (Other); University of Cambridge (Other); CURED Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-3521
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-11

CONDITIONS: Eosinophilic Esophagitis; EoE
Keywords: Eosinophilic Esophagitis; EoE; Cytosponge
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- EoE Patients (Experimental): Patients who have been diagnosed with EoE as per recent guidelines will be enrolled. Samples will be obtained using the Cytosponge™ Cell Collection Device (Cytosponge) prior to participants' routine endoscopy with biopsy.
  Interventions: Device: Cytosponge™ Cell Collection Device

INTERVENTIONS:
Device: Cytosponge™ Cell Collection Device — The Cytosponge™ Cell Collection Device (Cytosponge) is intended to collect surface cells from the esophagus. The device consists of a swallowable capsule, which dissolves in the body cavity, releasing a self-expandable sponge. The sponge is then retrieved from the esophagus using an attached cord. During the retrieval process, the sponge collects cells from the most superficial layer of the esophageal mucosa. Once removed from the body cavity, the sponge and cells are retained for investigation and/or testing. The Cytosponge™ Cell Collection Device (Cytosponge) received 510(k) clearance from the FDA on November 26, 2014 (K142695). The Cytosponge ™ Cell Collection device is a Class II product under 21 CFR 874.4710 esophagoscope (flexible or rigid) and accessories.
  Other Names: Cytosponge

SUMMARY:
The current endoscopic methods for diagnosing and monitoring treatment response in Eosinophilic Esophagitis (EoE) are costly, inconvenient, and risky. Novel diagnostic methods are needed, and the minimally-invasive Cytosponge holds great promise. It has been shown to be safe and accurate in Barrett's esophagus, it has the advantage (over the string test) of obtaining a true tissue sample, and our preliminary data supports its further study in EoE. The proposed prospective cohort study, conducted by experts in esophageal diseases and EoE, will assess the accuracy of Cytosponge compared to endoscopy and biopsy in EoE, and determine the safety and acceptability of this technique. Use of the Cytosponge would fundamentally change the paradigm for clinical management of EoE by allowing collection of non-endoscopic esophageal biopsies, thus minimizing the need for invasive testing. It would also facilitate future genetic, mechanistic, and pathogenesis research in EoE.

DETAILED DESCRIPTION:
Study design overview (all Aims) This will be a prospective cohort study, with patient enrollment conducted at UNC and Mayo Clinic with sample analysis performed by the University of Cambridge. In Aim 1, patients with EoE will be enrolled, tissue will be obtained from both the Cytosponge and endoscopy, and the methods will be compared for a single time point to determine accuracy of Cytosponge for quantifying esophageal eosinophil counts. For all patients, safety will be monitored and subjects will complete a survey about the acceptability of Cytosponge (Aim 2).

Cytosponge protocol:

After the study has been explained and a patient provides informed consent, the Cytosponge will be administered prior to endoscopy by trained research staff under physician supervision. If subjects opt to receive a local anesthetic, then they will be provided with a 2% lidocaine gargle prior to administration of the Cytosponge. The Cytosponge will be administered according to it's instructions for use. After retrieval, the string is cut and the sponge (which contains the tissue specimen) is placed in a container, immersed in fixative, and stored in a refrigerator at 4°C. The fixative is then spun in a centrifuge, and the pelleted cells are embedded in a paraffin block using standard techniques.

Upper endoscopy and biopsy:

After the Cytosponge has been removed, the patient will undergo standard of care (routine care) upper endoscopy and biopsy, as clinically indicated. During this exam, research staff will record all endoscopic features of EoE, including rings, furrows, white plaques, decreased vascularity, and strictures. The severity of the endoscopy findings will be measured using the recently validated endoscopic reference score (EREFS) scoring system. Four esophageal biopsies will be taken both from the distal (5 cm above the gastro-esophageal junction) and proximal (15 cm above the gastro-esophageal junction) esophagus. This number of biopsies has been shown to maximize the diagnostic sensitivity for EoE.

Histology and eosinophil counts:

All tissue samples from the Cytosponge and endoscopy will be coded with a subject's identification number, but will otherwise be masked for all clinical data, including EoE activity, symptoms, patient characteristics, and treatments prescribed. Using the paraffin blocks, pathology slides will be cut and the tissue processed with routine H&E staining. The slides will then be digitized, and using the Aperio ImageScope (Aperio Technologies, Vista, CA), the maximum eosinophil density (eosinophils/mm2 [eos/mm2]) will be determined using our previously validated protocol. For purposes of comparison to previous studies, eosinophil density will then be converted to eosinophil counts (eos/hpf) for an assumed hpf size of 0.24 mm2, the size of an average field as reported in the literature. The study pathologists from UNC and Mayo Clinic will review the specimens from their sites, and the study pathology from Cambridge will provide a second review of all specimens to ensure the most accurate quantification of eosinophil counts possible.

In addition, investigators plan to perform special staining and analysis of the existing biopsy and sponge samples with the goal of determining if the diagnostic accuracy of this test can be improved. In particular investigators will examine markers of eosinophil function, activation, and inflammation, such as eosinophil peroxidase (EPX), a granule protein that clearly identifies intact eosinophils, as well as extracellular EPX deposition suggestive of degranulation. This can be detected with immunohistochemistry. This would be done at Mayo clinic with our current collaborators who currently have the coded specimens.

Safety and accessibility assessments:

Patients will be assessed at multiple points to determine the safety of the Cytosponge in EoE. Investigators will assess for any symptoms or events as soon as the sponge capsule is swallowed, as well as immediately after the expanded sponge is removed. Participants will be contacted 1 and 7 days after the endoscopy to assess for adverse events. For Aim 2, participants will be administered the acceptability survey at the 7 day follow-up point, so patients have adequate time to reflect on their experiences with both tissue collection approaches. In particular this survey will record the patient's experience with swallowing the Cytosponge, whether they would do it again, and whether they prefer the Cytosponge or endoscopy for diagnosis and monitoring of EoE.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, comprehend, and complete the informed consent form
* Male or female subjects, age 18-80 years,
* Suspected EoE or has a diagnoses of EoE with current active disease,

Exclusion Criteria:

* History of esophageal stricture precluding passage of the endoscope or sponge,
* Pregnancy, or planned pregnancy during the course of the study,
* Any history of esophageal varices, liver impairment of moderate or worse severity (Child's- Pugh class B & C) or evidence of varices noted on any past endoscopy,
* Any history of esophageal surgery, except for uncomplicated fundoplication
* History of coagulopathy, with international normalized ratio (INR) >1.3 and/or platelet count of <75,000.
* Current use of blood thinners such as coumadin, warfarin, clopidogrel, heparin and/or low molecular weight heparin (requires discontinuation of medication 7 days prior to and 7 days after esophagogastroduodenoscopy (EGD) and Cytosponge administration, aspirin use is OK).
* Are allergic to local anesthetics such as lidocaine (these subjects may opt not to receive the optional lidocaine gargle prior to the Cytosponge administration and still be eligible).
* Have not fasted the night before administration of the Cytosponge.
* History of perforation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Dellon, MD, MPH, Principal Investigator — UNC-Chapel Hill
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirano I, Moy N, Heckman MG, Thomas CS, Gonsalves N, Achem SR. Endoscopic assessment of the oesophageal features of eosinophilic oesophagitis: validation of a novel classification and grading system. Gut. 2013 Apr;62(4):489-95. doi: 10.1136/gutjnl-2011-301817. Epub 2012 May 22. PMID 22619364
- [Background] Gonsalves N, Policarpio-Nicolas M, Zhang Q, Rao MS, Hirano I. Histopathologic variability and endoscopic correlates in adults with eosinophilic esophagitis. Gastrointest Endosc. 2006 Sep;64(3):313-9. doi: 10.1016/j.gie.2006.04.037. PMID 16923475
- [Background] Dellon ES, Fritchie KJ, Rubinas TC, Woosley JT, Shaheen NJ. Inter- and intraobserver reliability and validation of a new method for determination of eosinophil counts in patients with esophageal eosinophilia. Dig Dis Sci. 2010 Jul;55(7):1940-9. doi: 10.1007/s10620-009-1005-z. Epub 2009 Oct 15. PMID 19830560
- [Background] Dellon ES, Aderoju A, Woosley JT, Sandler RS, Shaheen NJ. Variability in diagnostic criteria for eosinophilic esophagitis: a systematic review. Am J Gastroenterol. 2007 Oct;102(10):2300-13. doi: 10.1111/j.1572-0241.2007.01396.x. Epub 2007 Jul 7. PMID 17617209
- [Result] Katzka DA, Smyrk TC, Alexander JA, Geno DM, Beitia RA, Chang AO, Shaheen NJ, Fitzgerald RC, Dellon ES. Accuracy and Safety of the Cytosponge for Assessing Histologic Activity in Eosinophilic Esophagitis: A Two-Center Study. Am J Gastroenterol. 2017 Oct;112(10):1538-1544. doi: 10.1038/ajg.2017.244. Epub 2017 Aug 15. PMID 28809387

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EoE Patients
Started | 86
Completed | 80
Not Completed | 6
Not completed — Unable to swallow Cytosponge | 6

BASELINE CHARACTERISTICS:
Population: Baseline characteristics unavailable for the 6 participants who were unable to swallow the Cytosponge.
Arm/Group | EoE Patients
Number analyzed (Participants) | 80
Age, Continuous [Mean (Full Range); unit: years] | 42 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 80
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Percent Agreement Between Cytosponge and Endoscopic Biopsy Results
Description: The primary outcome variables are sensitivity (percent agreement between positive results) and specificity (percent agreement between negative results) of the Cytosponge ability to detect the presence of EoE as compared to upper endoscopy with biopsy (the gold standard for diagnosis and monitoring of EoE). Overall agreement is defined as percentage of Cytosponge procedures yielding results consistent with endoscopic biopsy results. Presence of EoE is measured by the count of eosinophils present per high power field (eos/HPF) with active EoE defined as >=15 eos/HPF.
  Sensitivity was calculated via percentage of positive (active EoE) results obtained via Cytosponge as compared to results indicating active EoE via endoscopy with biopsy.
  Specificity was calculated via percentage of negative (inactive EoE) results obtained via Cytosponge as compared to results indicating inactive EoE via endoscopy with biopsy.
Time Frame: At study enrollment and initial procedure and each additional procedure, up to 1 year after enrollment
Population: Of the 105 procedures performed on 80 participants, 101 yielded results from both Cytosponge and endoscopy with biopsy for comparison.
Measure: Number; unit: Percent
Units Other Than Participants: Evaluable Specimens
Arm/Group | EoE Patients
Number analyzed (Participants) | 80
Number analyzed (Evaluable Specimens) | 101
Percent
  Sensitivity | 75
  Specificity | 86
  Overall Agreement | 80

2. Secondary Outcome: Overall Agreement Between Cytosponge and Endoscopic Biopsy Results as Measured by Kappa
Description: Overall agreement (Cytosponge procedures yielding results consistent with endoscopic biopsy results) as measured by Cohen's Kappa. Overall Cohen's Kappa is a statistical measure for assessing the reliability of agreement between the two results by taking into account the element of chance. Cohen's kappa can range from 0 to 1 with 1 indicating perfect agreement and 0 indicating an agreement equivalent to chance.
Time Frame: At study enrollment and initial procedure and each additional procedure, up to 1 year after enrollment
Population: Of the 105 procedures performed on 80 participants, 101 yielded evaluable specimens from both Cytosponge and endoscopy with biopsy for comparison.
Measure: Number; unit: Kappa coefficient
Units Other Than Participants: Results of Evaluable Specimens
Arm/Group | EoE Patients
Number analyzed (Participants) | 80
Number analyzed (Results of Evaluable Specimens) | 101
Kappa coefficient | 0.61
Statistical Analysis 1: Comparison: EoE Patients; All participants enrolled (EoE Patients) provided both a Cytosponge specimen and endoscopic biopsy. The results of these specimens were compared to examine overall agreement; Test type: Other — Overall agreement was calculated using Cohen's Kappa, with endoscopic biopsy as the gold standard; p = 0.0001, Cohen's Kappa — A p-value of <0.05 was considered statistically significant

3. Secondary Outcome: Acceptability of Cytosponge Compared to Endoscopic Biopsy, as Measured by Visual Analog Scale
Description: Acceptability of Cytosponge compared to endoscopic biopsy as measured by visual analogue scale. Participants were asked to rate their experience of the procedures on a scale of 0-10, where 0 indicates "unacceptable, very difficult even for a medical test," and 10 indicates "not an issue, would take test." A higher score indicates a more acceptable test. Acceptability was measured after each procedure and scores from each assessment were summed to obtain the mean and standard deviation.
Time Frame: 7 days after each procedure
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EoE Patients
Number analyzed (Participants) | 80
Units on a scale
  Cytosponge Acceptability | 7.24 (2.21)
  Endoscopy with Biopsy Acceptability | 5.83 (2.90)

4. Secondary Outcome: Acceptability of Cytosponge as Measured by the Impact of Events Scale
Description: Acceptability of Cytosponge as measured by the Impact of Events (IES) scale. The IES measures subjective distress (such as intrusive thoughts or emotions and avoidant or anxious behavior) following a stressful event. Respondents are asked to answer questions to indicate the amount of stress from the event.
  Scores are calculated using the following scale: Not at all =0, Rarely =1, Sometimes =3, Often =4. The total score is calculated by adding each response, with a total final score ranging from (0-60). Scores ranging 0-8 indicate no meaningful impact, scores ranging 9-25 indicate impact, and scores of 26 and above are considered very important (26-43 = powerful impact, 44-75 = severe impact).
  Acceptability was measured after each procedure and scores from each assessment were summed to obtain the mean and standard deviation.
Time Frame: 7 days after each procedure
Population: Not all participants competed the IES scale. Mean and Standard Deviation are reported for the 18 participants who completed the IES scale seven days after the procedure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | EoE Patients
Number analyzed (Participants) | 18
Units on a scale | 1.4 (2.7)

5. Other Pre Specified Outcome: Number of Responses Indicating Preference for Cytosponge Over Endoscopic Biopsy
Description: The number of responses indicating preference for Cytosponge to endoscopic biopsy. Preference was measured by asking participants after each procedure, "which procedure would you prefer to undergo again if your physician indicated it was medically necessary?" with the options "Traditional Upper Endoscopy" and "Cytosponge." The total number of responses recorded as "Cytosponge" and the total number of responses recorded as "Traditional Upper Endoscopy" were summed.
Time Frame: 7 days after each procedure
Population: Data reported for participants who indicated a preference at follow up.
Measure: Number; unit: responses
Arm/Group | EoE Patients
Number analyzed (Participants) | 48
responses
  Cytosponge Preferred | 42
  Endscopic Biopsy Preferred | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each procedure (interventional procedure and specimen collection) through 30-days post-procedure, up to 1 year
Description: Per study protocol section 7.2, only those events that are potentially related to participation in this research study were collected.
Arm/Group | EoE Patients
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 0/86

LIMITATIONS AND CAVEATS:
Due to device availability, this study was suspended indefinitely in June 2016. In August 2020, the decision was made to terminate the study early. The study population was limited to adult patients without critical strictures or small caliber esophagus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02114606/Prot_SAP_000.pdf